CLINICAL TRIAL: NCT03420729
Title: Acceptability and Tolerability of Magnetic Assisted Capsule Endoscopy Compared to Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STH19595
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Gastroscopy; Endoscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnetic assisted capsule endoscopy (Experimental): All participants will undergo magnetic assisted capsule endoscopy at the sloan medical centre
  Interventions: Procedure: gastroscopy; Device: magnetic assisted capsule endoscopy
- gastroscopy (Active Comparator): All participants will undergo gastroscopy as standard of care at sheffield teaching hospitals
  Interventions: Procedure: gastroscopy; Device: magnetic assisted capsule endoscopy

INTERVENTIONS:
Procedure: gastroscopy — a thin, flexible tube called an end oscope is used to look inside the oesophagus (gullet), stomach and first part of the small intestine (duodenum)
Device: magnetic assisted capsule endoscopy — The patient will be given 500 to 1000mls of water with 6 drops of simethicone added to drink. This is to enable adequate distension of the stomach. The patient then swallows the capsule in the presence of the PI. MACE of the oesophagus and stomach will be carried out by the PI. Once the PI is satisfied that an adequate examination has been completed the capsule will be allowed to pass into and through the small bowel.

SUMMARY:
Dyspepsia is a common presenting complaint that doctors have to manage and this is true both in the primary and secondary care setting. OGD is a useful test for investigating a variety of suspected upper GI disorders including dyspepsia. However, it is uncomfortable for patients and incurs the risk of intubation and sedation. Capsule endoscopy (CE) is the investigation of choice for diseases of the small bowel. It is safe, non-invasive and well tolerated, the main risk being capsule retention occurring in up to 1-2% of procedures.

The investigators wish to undertake a prospective study comparing acceptability and tolerability of MACE and OGD in the investigation of dyspepsia. Patients presenting to general practice or the outpatients department with symptoms of dyspepsia who are referred for investigation are invited to take part in the study. Patients will undergo MACE prior to OGD performed by an endoscopist blinded to the MACE findings. . A comparison of tolerance and acceptance of both procedures will be measured by means of using structured and validated, qualitative questionnaires. The aim is to assess for whether there is a significant difference between the perception and experience of both modalities.

DETAILED DESCRIPTION:
This is a prospective, single blinded, comparative trial of patient acceptability and tolerability of MACE and both transoral and transnasal gastroscopy in the investigation of dyspepsia.

The study will be conducted within Sheffield Teaching Hospitals. Recruitment will take place at the Sloan Medical Centre, the Royal Hallamshire Hospital or the Northern General Hospital during the consultation when patients present with dyspepsia requiring gastroscopy for investigation as per national guidelines. MACE will take place at the Sloan Medical Centre. Equipment for collecting demographics (height, weight etc) will be available. All the capsule equipment is stored and re-charged in this designated room. The case report files and computer data will be stored in this room that is secured by a locked door.

Gastroscopy will take place in the Endoscopy Departments, which are specially designed units for a variety of endoscopic tests, at the Royal Hallamshire Hospital and Northern General Hospital.

Patients are assessed in the Sloan Medical Centre or the Royal Hallamshire Hospital/Northern General Hospital outpatients department for their primary presenting complaints of dyspepsia. The study will be discussed with patients in those who satisfy the enrolment criteria and they will be provided by with the written study literature. If in agreement to enter the study, informed written consent will be obtained from the patient.

Prior to any investigation, the pre-MACE section of the questionnaire will be completed by the patient with the assistance of study team members. MACE will be performed at the Sloan Medical Centre; this will be in a dedicated room setup to accommodate the MACE procedure.The post-MACE section of the questionnaire will then be completed by the patient with the assistance of study team members. MACE will be preceded by obtaining measurements of height, weight and waist/hip circumference. The patient will then be given 500 to 1000mls of water with 6 drops of simethicone added to drink. This is to enable adequate distension of the stomach. Our previous study has shown excellent tolerance of this volume of water distension by patient.

The patient then swallows the capsule in the presence of the PI. MACE of the oesophagus and stomach will be carried out by the PI. Once the PI is satisfied that an adequate examination has been completed the capsule will be allowed to pass into and through the small bowel. Visibility of major locations of the stomach will be documented. Any pathology noted will be recorded according to the standard fashion described for gastroscopy reporting. A note of the procedure duration will be recorded. The patient will be given the option to complete their small bowel capsule endoscopy in the standard way and this will be reported in the usual fashion.

Patients referred for gastroscopy as part of the normal pathway for investigation of dyspepsia, will attend a designated list for their gastroscopy within 1 week and this will be performed by a JAG accredited endoscopist who has experience in endoscopic therapy. TOG will be performed using a standard 11mm Olympus or Pentax gastroscope and TNG will be performed using an ultra-thin 5.9mm Olympus or Fujinon gastroscope. The endoscopist performing the gastroscopy will be a member of the study team. The participant will be asked to complete the pre-gastroscopy section of the participant questionnaire before, and the post-gastroscopy section after the procedure.

Patients will have 80mg simethicone mixed in 100mls of water as an anti-foaming agent prior to the gastroscopy. Patients undergoing TNG will have their nasal passages prepared with a fine mist of 5% lidocaine and 0.5% phenylephrine (co-phenylephrine nasal spray) which are a local anaesthetic and nasal decongestant. Phenylephrine is a topical vasoconstrictor used as a nasal decongestant to reduce the risk of peri-procedure epistaxis. Five minutes following this, a 6mm diameter soft-sillicone catheter lubricated with 2% aqueous lidocaine gel is inserted into either or each nasal passage approximately 5-8cm passages to ensure the passage is wide enough to comfortably accommodate a nasal endoscopy. If neither passages accommodate the silicone catheter, the procedure will be converted to a transoral route. Patients undergoing TOG will have 10 sprays of 10% topical lidocaine administered to the oropharynx. Procedures will be performed in the left lateral decubitus position.

Gastroscopy will be performed in the standard fashion and reported to the PI to compose a written record for study purposes. This reporting system (InfoFlex) requires details to be entered regarding indication for examination, patient comfort, sedation and pathology. Pathology will be documented in a standardised way (for further details see section on Scientific Justification). An entry of the duration of procedure will be included. This denotes the end of the participants' involvement in the study. The patient will be managed thereafter according to the responsible clinician at the Sloan Medical Centre or Sheffield Teaching Hospitals NHS Trust.

The primary outcome will be evaluated using the questionnaires to compare acceptability and tolerance of both procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over and up to but not exceeding 80 years
* Patients presenting symptoms of dyspepsia whom require gastroscopy as per national guidelines

Exclusion Criteria:

Patients under the age of 18 years

* Patients over the age of 80 years
* Active vomiting
* Patients with a permanent pacemaker, implantable cardioverter-defibrillator or REVEAL device
* Patients with any electronic/magnetic/mechanically controlled devices e.g. sacral nerve stimulators, bladder stimulators
* Patients with dysphagia, odynophagia or known swallowing disorder
* Patients with known Zenker's diverticulum
* Patients with suspected bowel obstruction or bowel perforation
* Patients with prior bowel obstruction
* Patients with gastroparesis or known gastric outlet obstruction
* Patients with known Crohn's disease
* Patients who are taking daily non-steroidal anti-inflammatory drugs (excluding prophylactic doses of aspirin) for more than six months
* Patients who have received abdominopelvic radiotherapy treatment
* Patients with a history of GI tract surgery (Billroth I, Billroth II, Oesophagectomy, gastrectomy or bariatric procedure)
* Patients that are pregnant or lactating
* Patients with altered mental status that would limit their ability to swallow
* Patients with allergy to conscious sedation or metoclopramide
* Patients unwilling to swallow the capsule
* Patients with known dementia affecting ability to consent
* Patients who are unable to understand or speak English
* Patients unable to provide written informed consent
* Patients with head and neck cancers
* Patients who have had nasal surgery, eg. rhinnoplasty
* Patients allergic to lidocaine, pheylephirine or midazolam
* Patient with bleeding diathesis, on warfarin or have chronic liver disease
* Patients reluctant to have gastroscopy by both oral or transnasal route

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Endoscopy Concerns Score | procedure
  Differences in the Endoscopy Concerns Score (ECS) when patients have magnetic assisted capsule endoscopy (MACE) and when they have conventional gastroscopy

SECONDARY OUTCOMES:
Clinician rating of visualization of upper GI Tract | procedure
  Differences in visualization of the upper GI tract

CONTACTS AND LOCATIONS:
Overall Officials: Mark McAlindon, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom